CLINICAL TRIAL: NCT01077063
Title: An Early Safety and Efficacy Study of Ascites Management: Standard Paracentesis or Early Intervention With Pleurx Catheters in Patients With Malignant Ascites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed by PI because of low enrollment.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0940; Carefusion (Other Grant/Funding Number: Carefusion)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Malignant Ascites
Keywords: Pleurx catheter; malignant ascites
MeSH Terms: interventions — Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paracentesis (Active Comparator): cutting and draining procedure for malignant ascites
  Interventions: Procedure: paracentesis
- Pleurx catheter (Active Comparator): a catheter drainage system the subject uses himself/herself.
  Interventions: Device: Pleurx catheter

INTERVENTIONS:
Procedure: paracentesis — surgical drainage of malignant ascites
  Arms: paracentesis
Device: Pleurx catheter — take home catheter drainage system that the subject uses himself/herself as needed.
  Arms: Pleurx catheter

SUMMARY:
The purpose of this study is to assess in a controlled prospective setting, the safety of the use of Pleurx catheters and standard therapeutic paracentesis in patients with malignant ascites.

DETAILED DESCRIPTION:
Study Design: Single institution, open-label, randomized study

Study Device: Pleurx Catheter

Treatment Plan: Cohort A: 15 patients treated with standard therapy (therapeutic paracentesis +/- diuretics)

Cohort B: 15 patients treated with peritoneal Pleurx catheter

Duration of Participation: Patients will be followed for one year, or until death, whichever comes first.

Primary Outcome: Safety of the Pleurx catheter procedure or paracentesis

Secondary outcomes: Overall complications, quality of life, overall survival, and symptom control

ELIGIBILITY:
Inclusion Criteria:

(Patients can receive chemotherapy at the discretion of treating oncologist)

1. Patients with recurrent malignant ascites
2. Patients with refractory malignant ascites
3. Proven malignancy
4. Age >= 18 years old
5. Eastern Cooperative Oncology Group (ECOG) performance scale =< 2
6. Ability to understand and willingness to sign a written informed consent

Definitions:

Malignant ascites: One of the following criteria

1. Positive ascitic fluid cytology
2. Histology proven malignancy with imaging studies with evidence of liver metastasis and ascites
3. Malignant Budd Chiari Syndrome with associated ascites
4. Hepatocellular carcinoma and ascites
5. Chylous ascites due to lymphoma
6. Peritoneal carcinomatosis and concurrent ascites
7. Proven abdominal malignancy with concurrent ascites

Refractory / Recurrent ascites: One of the following criteria

1. Symptomatic ascites that recurred after one paracentesis in a patient with known malignant ascites.
2. Symptomatic ascites that did not respond clinically to at least two weeks of diuretics. Use of diuretics at the discretion of the treating physician.
3. Intolerance or relative contraindications to diuretics: (serum sodium (Na) concentration of <125 mmol per liter or serum creatinine >1.5 mg/dl, hyperkalemia (potassium >5.2 mEq/L or azotemia Bun/Creatinine ratio > 20).
4. Removal of at least 5 L in the preceding two months for symptoms relief

Exclusion criteria:

1. Life expectancy less than one month
2. Coagulopathy (international normalized ratio [INR] > 2 that does not correct with fresh frozen plasma)
3. Hepatorenal syndrome
4. Active skin infections at abdomen before procedures
5. Inability to provide inform consent
6. Platelet counts < 50,000/mcL
7. Uncontrolled illness including, but not limited to, ongoing or active infection requiring intravenous (IV) antibiotics, that the physician feels would increase the risk of infection with the procedures or white blood cell (WBC) count > 20,000/mcL
8. Absolute neutrophil count <1000 / cu mm
9. Pregnant women
10. Multiloculated ascites

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pleurx Catheter | Paracentesis
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: subjects with malignant ascites
Groups:
- Total: Total of all reporting groups
Arm/Group | Paracentesis | Pleurx Catheter | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 53.67 [42 to 62] | 55 [45 to 70] | 54.42 [42 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety of Pleurx Catheter or Paracentesis
Description: Primary Outcome: Safety of the Pleurx catheter procedure or paracentesis
  Safety of the pleurx catheter procedure or paracentesis. Safety will be assessed by the degree of unacceptable toxicities, defined as life threatening complications related to the procedure. These include peritonitis, perforation, or death related to the procedure.
Time Frame: 3 years
Measure: Number; unit: events
Arm/Group | Paracentesis | Pleurx Catheter
Number analyzed (Participants) | 3 | 4
events
  Related peritonitis | 0 | 0
  Related death | 0 | 0
  Related perforation | 0 | 0
  Unnacceptable other (related) | 0 | 1

ADVERSE EVENTS:
Arm/Group | Paracentesis | Pleurx Catheter
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracentesis (N=3) | Pleurx Catheter (N=4)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
infection (non septic) (Infections and infestations) | 0 (0) | 1 (1)
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
peritonitis (Infections and infestations) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracentesis (N=3) | Pleurx Catheter (N=4)
↑ alkaline phosphatase (Investigations) | 1 (2) | 3 (4)
↑ ALT (Investigations) | 2 (3) | 2 (4)
↑ AST (Investigations) | 1 (2) | 2 (3)
↑ CK serum (Investigations) | 1 (1) | 0 (0)
↑ creatinine (Investigations) | 1 (1) | 1 (1)
↑ glucose (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
↑ potassium (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
↑ magnesium (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
↑ total bilirubin (Investigations) | 1 (2) | 2 (2)
↑ PT (Investigations) | 0 (0) | 1 (1)
↑ PTT (Investigations) | 0 (0) | 2 (2)
↑ uric acid (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
↓ albumin (Metabolism and nutrition disorders) | 1 (3) | 2 (4)
↓ calcium (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
↓ glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
↓ hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 2 (5)
↓ lymphocytes (Blood and lymphatic system disorders) | 2 (6) | 2 (3)
↓ magnesium (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
↓ sodium (Metabolism and nutrition disorders) | 2 (3) | 2 (5)
↓ platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
↓ potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
↓ total protein (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
↓ white blood cells (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (5)
anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
bilateral lower extremity pitting edema (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
dark urine (Renal and urinary disorders) | 0 (0) | 1 (1)
daytime somnolence (Nervous system disorders) | 0 (0) | 1 (1)
decreased appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
early satiety (Gastrointestinal disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (4) | 1 (2)
icterus (General disorders) | 0 (0) | 1 (1)
loss of muscle mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1) | 1 (2)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
numbness right foot (Nervous system disorders) | 1 (1) | 0 (0)
rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
reddened rash on abdomen (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed by investigator due to low enrollment. Subject JH006 S-B did have abdominal pain, post Pleurx placement, so it was removed and she was taken out of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes